CLINICAL TRIAL: NCT02771171
Title: Volumetric Three-dimensional Analysis of the Pediatric Upper Airway Shape Using Computed Tomography Imaging.
Status: Completed | Type: Observational
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Tariq Wani, Consultant Anesthesiologist, King Fahad Medical City
Other Study IDs: IRB
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Airway Management
Keywords: Pediatric Airway, Three-dimensional Imaging, CT Scan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Age groups: The cohort is divided into on the basis of age
  Interventions: Radiation: CT Scan

INTERVENTIONS:
Radiation: CT Scan — CT imaging

SUMMARY:
CT and MRI based measurements of the pediatric airway has changed the age-old cone shape concept of the pediatric airway and define airway shape as elliptical structure. The cone shape was based on the cadaveric measurements done by Bayeux in 1897 and described later by Eckenhoff in 1951.

The present study is based on three-dimensional CT images of the airway column replicating the cylinders used by Bayeux for his cadaveric measurements. The purpose of this study was to determine the cone shape of the pediatric airway.

DETAILED DESCRIPTION:
This is a retrospective review of three-dimensional CT air column images of 60 children aged 1 month to 8 years undergoing radiological evaluation unrelated to airways symptomatology. The CT scans will be evaluated in children either sleeping naturally or sedated throughout the study period. Volumetric analysis of the air-column was done at the level of cricoid, subglottis and trachea

Exclusion Criteria:

Patients with a tracheostomy or endotracheal tube in place, tracheo-esophageal fistula, pulmonary collapse or atelectasis, mediastinal mass, diaphragmatic hernia, extrapulmonary and intrathoracic mass, preterm infants, and patients with genetic syndromes and primary lung diseases.

Patients with poor image quality were also excluded from the study.

ELIGIBILITY:
Inclusion Criteria: Children aged 1 month to 96 months

Exclusion Criteria:

Patients with a tracheostomy or endotracheal tube in place, tracheo-esophageal fistula, pulmonary collapse or atelectasis, mediastinal mass, diaphragmatic hernia, extrapulmonary and intrathoracic mass, preterm infants, and patients with genetic syndromes and primary lung diseases Patients with poor image quality were also excluded from the study.

Ages: 1 Month to 96 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1 month to 8 years undergoing radiological evaluation (CT Imaging) unrelated to airways symptomatology
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Shape of the pediatric Airway | 12 months
  The purpose of this study was to determine the shape of pediatric airway from subglottis to the trachea using 3D dimensional CT air column images. The shape of the airway was calculated on the basis of the volumes of airway column at the level of subglottis, cricoid and trachea

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tobias, MD, Study Director — Nationwide Children's Hospital, Columbus, Ohio
Locations (1):
- King Fahad Medical City, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] ECKENHOFF JE. Some anatomic considerations of the infant larynx influencing endotracheal anesthesia. Anesthesiology. 1951 Jul;12(4):401-10. doi: 10.1097/00000542-195107000-00001. No abstract available. PMID 14847223
- [Result] Wani TM, Bissonnette B, Rafiq Malik M, Hayes D Jr, Ramesh AS, Al Sohaibani M, Tobias JD. Age-based analysis of pediatric upper airway dimensions using computed tomography imaging. Pediatr Pulmonol. 2016 Mar;51(3):267-71. doi: 10.1002/ppul.23232. Epub 2015 Jun 17. PMID 26083203
- [Result] Litman RS, Weissend EE, Shibata D, Westesson PL. Developmental changes of laryngeal dimensions in unparalyzed, sedated children. Anesthesiology. 2003 Jan;98(1):41-5. doi: 10.1097/00000542-200301000-00010. PMID 12502977